CLINICAL TRIAL: NCT02800174
Title: Use of the Smart Nitinol Stent System for the Treatment of Severe Atherosclerotic Carotid Stenosis: Study Protocol for a Retrospective, Non-randomized, Long-term Parallel Controlled Trial
Brief Title: Smart Nitinol Stent System for the Treatment of Severe Atherosclerotic Carotid Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, Zhigang Ma, Director, Beijing Jishuitan Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BeijingJH_001
Record Dates: First submitted 2016-06-12; First posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Carotid Artery Stenosis
MeSH Terms: conditions — Carotid Stenosis | interventions — Platelet Aggregation Inhibitors; Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Smart nitinol stent implantation group (Experimental): The Smart nitinol stent system was used (import product registration number YZB/USA 0115-2008; Nitinol stent system, trade name SMART Control). The stent system comprises a self-expanding stent and a delivery system. The self-expanding stent is composed of a nickel titanium alloy and the ends of the stent are equipped with tantalum radiopaque markers. The Smart nitinol stent system is sterilized with ethylene oxide gas and is intended for single use only.
  Interventions: Device: Smart nitinol stent implantation
- Antiplatelet drug group (Active Comparator): Patients with carotid artery stenosis treated conservatively were commenced on an indefinite course of one or more oral antiplatelet drugs. The antiplatelet regimes comprised 100 mg or 300 mg aspirin before sleep with clopidogrel 125 mg or 250 mg daily; or 75 mg clopidogrel before sleep daily.
  Interventions: Drug: antiplatelet drug

INTERVENTIONS:
Device: Smart nitinol stent implantation — Before intervention, clopidogrel (75 mg/d), aspirin (100 mg/d) and atorvastatin (40 mg/d) were prescribed. One week later, aortic arch and aortocranial angiography were performed under general anesthesia to determine the site, range and extent of the lesion and the status of the cerebral microcirculation, and consequently to inform the treatment strategy and the selection of the correct size of self-expanding nitinol stent system.
  Arms: Smart nitinol stent implantation group
Drug: antiplatelet drug — Patients with carotid artery stenosis treated conservatively were commenced on an indefinite course of one or more oral antiplatelet drugs. The antiplatelet regimes comprised 100 mg or 300 mg aspirin before sleep with clopidogrel 125 mg or 250 mg daily; or 75 mg clopidogrel before sleep daily.
  Other Names: aspirin and clopidogrel
  Arms: Antiplatelet drug group

SUMMARY:
To validate the long-term effects of implantation of the self-expanding Smart nitinol stent system for the treatment of severe atherosclerotic carotid stenosis in a 2-year follow-up study of a large patient cohort

DETAILED DESCRIPTION:
Atherosclerosis is a leading cause of carotid artery stenosis. The risk of atherosclerosis increases with age, occurring mainly in middle-aged and elderly populations. The morbidity and mortality of stroke caused by atherosclerosis also increase with aging. An epidemiologic study demonstrated that carotid artery intima-media thickness is a marker of atherosclerotic peripheral arterial disease, and found evidence that the likelihood of a clinical diagnosis of atherosclerosis increases two- to threefold from 20 to 90 years of age. The risk of atherosclerosis also increases with age in animals fed atherosclerosis-inducing diets. The close relationship between atherosclerosis and aging shows that atherosclerosis is a chronic and progressive degenerative disease.

Atherosclerotic carotid stenosis is an independent risk factor for ischemic cerebrovascular disease. Vascular stenting of carotid artery stenosis is an increasingly popular technique. It is safe, quick, minimally invasive, can be performed under local anesthesia, and can be used to treat proximal and intracranial lesions. Vascular stenting enables flow to be restored in previously narrowed vessels, restoring blood supply to the brain and preventing plaque rupture. Carotid artery stenosis of 70%-90% is considered the highest risk for stroke, and is a compelling indication for stenting. The Smart stent system (Cordis Corporation, Miami, FL, USA) is a nitinol self-expanding stent that is soft, elastic, has uniform radial tension and is readily endothelialized.

Phatouros et al. treated four patients with carotid artery stenosis >70% using self-expanding Smart stents and <20% residual stenosis was achieved in all cases; no transient ischemic attacks or new strokes occurred during a follow up period of 6 months. Drescher et al. also used self-expanding Smart stents in 13 patients with severe carotid artery stenosis and found no complications during a 6-month follow-up period. Wholey et al. deployed stents to treat carotid artery stenosis in more than 500 patients, and found that the rates of neurologic complications and restenosis were decreased after application of either balloon-mounted or self-expanding stents. Three-year follow-up results have shown that balloon-mounted stents lead to better vessel patency than self-expanding stents, but that balloon-mounted stents are vulnerable to compression. Lownie et al. examined the efficacy of self-expanding Smart stents in 21 patients with severe symptomatic carotid artery stenosis (stenosis >70%) without angioplasty. All patients were followed up for an average period of 19 months. Self-expanding Smart stents improved vascular stenosis and blood flow without the need for balloons or adjunctive protection devices.

Zhao et al. used Smart stents to treat patients with carotid artery stenosis of >65%, and found the treatment safe and effective, while observing no severe complications. Li et al. treated patients with carotid bifurcation and origin stenosis of >50% with self-expanding Smart stents, and found that patients' neurologic function improved to different extents, and that there were no strokes or transient cerebral ischemic attacks during a subsequent period of 13-14 months. Chen et al. used self-expanding Smart stents to treat 48 patients with carotid artery stenosis of 75%-99%, achieving favorable clinical outcomes in 43 (89.6%), with no recurrence of stenosis during a relatively short follow-up period of 1-6 months, and few postoperative complications or sequelae.

In a cohort of 38 patients with extracranial artery (internal carotid artery outer segment, vertebral artery or subclavian artery) stenosis treated with Smart stents and followed up for an average of 18 months, satisfactory clinical outcomes were achieved in 33 (86.8%). These investigators also treated another cohort of 41 patients with carotid artery stenosis with Smart stents, and concluded that vascular Smart stent deployment is an effective and safe method for treating carotid artery stenosis.

No long-term or randomized controlled trial evidence regarding the use of the Smart nitinol stent system for the treatment of atherosclerotic carotid stenosis currently exists. This study is a non-randomized controlled trial, in which deployment of the Smart nitinol stent system will be compared with conservative management with platelet aggregation inhibitors in a group of patients with severe atherosclerotic carotid stenosis subsequently followed up for 2 years.

Adverse events Possible adverse events associated with Smart stent implantation include vascular spasm, bradycardia, hypotension, luxury perfusion syndrome, intraoperative thrombosis and thrombus detachment, ischemic stroke, intraoperative hypertension, postoperative hypotension and hypoglycemia. If adverse events occur, details of the event including the date of occurrence, measures taken related to the treatment, causal relationship with the treatment and treatment of the adverse event will be reported to the principal investigator and the institutional review board within 24 hours.

Data collection, management, analysis and open access All data will be collected in case report forms and collated. Collated data will be input into an electronic database using a double-data entry strategy by trained professional staff. Information accuracy will be checked when all recruited patients are followed up. The database will be locked by the researcher in charge and will not be altered. All information relating to this trial will be preserved by Beijing Jishuitan Hospital, China. The electronic database will be fully disclosed to a professional statistician for statistical analysis. Anonymized trial data will be published at www.figshare.com.

Statistical analysis Statistical analysis will be performed by a statistician blinded to grouping using SPSS 14.0 software. Normally distributed measurement data will be expressed as the mean ± standard deviation, and numeration data as the frequency. The two sample t-test or rank sum test will be used to compare the means of measurement data between the stent implantation and drug groups. The chi-squared test will be used to compare numeration data between the groups. Multivariate regression analysis will be used to compare mRS scores 2 years after treatment. Kaplan-Meier and Cox Proportional Hazards Survival regression analysis will be used to examine survival time and survival state. A P value <0.05 will be considered statistically significant.

Frequency and measures for monitoring trial implementation Trial progression will be reported to the ethics committee of Beijing Jishuitan Hospital, China every 6-12 months and the trial's status will be updated in the registration database.

Confidentiality principle The electronic database will be preserved in a dedicated password-protected computer and managed by a data management professional. Data recorded on paper will be preserved in a secure, locked place for future viewing.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Of either sex
* Carotid artery stenosis caused by atherosclerotic plaque
* Diagnosed with severe atherosclerotic carotid stenosis according to a previously described method (North American Symptomatic Carotid Endarterectomy Trial Collaborators, 1991)
* Severe carotid artery stenosis confirmed by transcranial Doppler and carotid duplex ultrasonography
* Provision of informed consent regarding trial procedure

Exclusion Criteria:

* Carotid artery stenosis caused by fibromuscular dysplasia, Takayasu's arteritis or radiation injury
* Severe central nervous system disorders, such as complete loss of cerebral function on the affected side with cerebral paralysis
* Life expectancy <2 years because of intracranial tumors or other diseases
* Pregnant or lactating
* Renal impairment (if use of contrast agent will worsen renal function)
* Concurrent hemorrhagic disease, or contraindication to antiplatelet or anticoagulant therapies for safety reasons
* Leakage of contrast agent indicative of vessel perforation
* Dilated aneurysm proximal or distal to stenotic foci
* Allergy to stent material
* Complete occlusion of the carotid artery or lesion length >10 mm, accompanied by intravascular thrombus and multiple segments of stenosis confirmed by imaging examination
* Intracranial hemorrhage within 3 weeks or large areas of cerebral infarction within 4 weeks of treatment
* Unable to or declined to cooperate with follow-up examination
* Unable to provide informed consent because of intellectual disability or language disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2006-06; Primary Completion 2007-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
mRS score | 2 years after treatment
  The mRS is a 7-point scale used to evaluate a patient's functional recovery.

SECONDARY OUTCOMES:
The recurrence of cerebrovascular events | 1 and 2 years after treatment
  The incidences of transient cerebral ischemia, cerebral infarction, cerebral hemorrhage or death because of cerebrovascular diseases will be recorded.
National Institute of Health stroke scale(NIHSS) score | 1 and 2 years after treatment
  The NIHSS is a 43-point scale, with higher scores indicative of more severe neurological deficits.

CONTACTS AND LOCATIONS:
Overall Officials: Zhigang Ma, Master, Principal Investigator — Beijing Jishuitan Hospital, China

IPD SHARING:
Plan to Share IPD: Undecided